CLINICAL TRIAL: NCT04544202
Title: Managed Access Program (MAP) Cohort Treatment Plan CDRB436F2001CM to Provide Access to Trametinib and Dabrafenib Combination Therapy in the Adjuvant Treatment of High-risk BRAF 600 Mutation-positive Melanoma After Surgical Resection
Brief Title: Compassionate Use Program BRAF Mutation-positive Patients in the Adjuvant Treatment of Melanoma After Surgical Resection
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436F2001CM
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Melanoma; Adjuvant
Keywords: Melanoma; Adjuvant; BRAF V600; Malignant skin cancer; Skin cancer; Stage III melanoma; Cutaneous; Resection; Surgical resection; Mutation; Compassionate Use; Dabrafenib; Trametinib; DRB436; TMT212; Cohort
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Dabrafenib and Trametinib — The starting dose of the combination treatment will be administered as follows:
  * Dabrafenib, 150 mg, twice daily (BID);
  * Trametinib, 2.0 mg, once daily (QD)
Drug: Dabrafenib — If administration of dabrafenib is interrupted or permanently discontinued, administration of trametinib may continue.
Drug: Trametinib — If administration of trametinib is interrupted or permanently discontinued, administration of dabrafenib may be continued.

SUMMARY:
The purpose of this Treatment Plan is to allow access to trametinib and dabrafenib for eligible high-risk BRAF mutation-positive patients in the adjuvant treatment of melanoma after surgical resection. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

DETAILED DESCRIPTION:
The requesting Treating Physician submitted a request for access to drug (often referred to as Compassionate Use) to Novartis which was reviewed and approved by the medical team experienced with the drug and indication.

This program will provide access to patients until:

* All participating countries have received marketing authorization and product is commercially available and accessible to all participating patient(s) or
* Alternative treatment options are available and/or
* In case of changes in the safety profile or a lack of overall efficacy of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Has or is willing to give consent to the Treating Physician in accordance with the local regulatory requirements.
2. Has the following diagnosis: Completely resected (R0) histologically confirmed high-risk (stage III) cutaneous melanoma with confirmed BRAF V600E/K activating mutation.

   Patients presenting with initial resectable lymph node recurrence after a diagnosis of Stage I or II melanoma are eligible. Patients with an unknown primary melanoma are not eligible.
3. All clinical trials that the patient might qualify for have been ruled out.
4. Is receiving care at a clinical site with a Treating Physician who has experience with administering investigational agents for patients with this condition, or the patient is willing and/or able to travel to a site and receive treatment under the guidance of physician with this experience.
5. Is able to retain oral medication and swallow tablets/capsules (appropriate exceptions allowed for patients who are unable to swallow tablets/capsules - this is subject to availability of alternative (liquid) oral formulations).
6. Is not eligible for participation in any of the IMP's ongoing clinical trials or has recently completed a clinical trial that has been terminated and, after considering other options (e.g., trial extensions, amendments, etc.), the clinical team has determined that treatment is necessary and there are no other feasible alternatives for the patient.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 3 (or equivalent) and is in stable clinical condition. NOTE: patient in rapidly deteriorating clinical condition prior to start of therapy should not be considered for this program.
8. Does not require treatment with prohibited concomitant medications (please refer to the IB or approved label/SmPC).
9. Women of childbearing potential must have had a negative serum β-human chorionic gonadotropin (HCG) pregnancy test within 7 days prior to starting dabrafenib and trametinib treatment. Subjects with a positive pregnancy test result must be excluded from the program. Subjects with a negative pregnancy test result must agree to use an effective contraception method as described below throughout the treatment period and for a total of 4 months following the last dose of treatment.

Contraceptive Methods for Females of Childbearing Potential:

* An intrauterine device with a documented failure rate of less than 1% per year
* Vasectomized partner who is sterile prior to the female patient's entry into the Compassionate Use program, and this male is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days prior to first dose of treatment, through the dosing period, and for at least 4 months after the last dose of treatment. Abstinence is only acceptable when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.
* Double-barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with vaginal spermicidal agent (foam/gel/cream/suppository).

Note: Hormonal-based methods (e.g., oral contraceptives) are not permitted as contraception due to potential drug-drug interactions with dabrafenib.

Females Not of Childbearing Potential Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) is defined as any female who has had a documented hysterectomy, bilateral oophorectomy (ovariectomy), bilateral tubal ligation or tubal occlusion, or is post-menopausal.

A practical definition accepts menopause after 1 year without menses with an appropriate clinical profile; e.g., age appropriate, >45 years in the absence of hormone replacement therapy (HRT). In questionable cases, the patient must have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value <40 pg/mL (<140 pmol/L).

Female patients determined not to be post-menopausal must use adequate contraception, as defined immediately above for females of childbearing potential.

Female subjects who are lactating must discontinue nursing prior to the first dose of program treatment and must refrain from nursing throughout the treatment period and for 4 months following the last dose of program treatment.

If a subject becomes pregnant during the treatment period of the program, the treatments should be stopped immediately.

Written patient informed consent must be obtained by the Treating Physician prior to start of treatment in accordance with the applicable local regulatory requirements.

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

History of hypersensitivity to any drugs or metabolites of similar chemical classes as the product.

1. Uveal or mucosal melanoma.
2. Evidence of metastatic disease.
3. Female who is pregnant or nursing (patient must discontinue nursing in order to enroll in the program).

   NOTE: Safety and efficacy in pregnant or nursing women has not been investigated. Inclusion of pregnant or nursing woman may be considered in individually upon review by the Novartis Country Pharma Organization Medical Advisor/Director.
4. Patients who have any lab abnormalities or AE/SAEs greater than Grade 3 (CTCAE v5.0)
5. Concurrent treatment with other systemic anti-cancer therapies is not allowed, with the exception of surgery (other exceptions might be allowed and are subject to individual evaluation). Patients who are currently being treated with another systemic anti-cancer therapy (e.g., chemotherapy, immune, biologic, or targeted therapy) must discontinue use prior to initiation of treatment with trametinib and dabrafenib. NOTE: Radiation skin injury has been reported with concurrent use of dabrafenib and radiation.
6. Presence of any malignancy with confirmed activating RAS mutation. NOTE: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.
7. Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or dabrafenib, or excipients or to dimethyl sulfoxide (DMSO).
8. Any medical conditions or physical examination or clinical laboratory findings which, would put the patient at high risk for an adverse outcome.
9. Current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy.
10. Current evidence of cardiovascular risk including any of the following:

    * LVEF<LLN
    * A QT interval corrected for heart rate using the Bazett's formula ≥ 480 msec
    * A clinically significant uncontrolled arrhythmias
    * Acute coronary syndrome (including myocardial infarction and unstable angina)
    * Congestive heart failure ≥ Class II as defined by New York Heart Association
11. Not able to understand and to comply with treatment instructions and requirements.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult